CLINICAL TRIAL: NCT04655274
Title: Comparision of Visual Outcomes and Patient Satisfaction Between Two Diffractive Trifocal Intraocular Lenses
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Aslı Çetinkaya Yaprak, Principal Investigator, Akdeniz University
Other Study IDs: 2020-11
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Cataract Senile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RayOne Trifocal intraocular lenses: Eyes of patients undergoing cataract surgery with implantation of RayOne Trifocal (Rayner IOL, Ltd.) intraocular lenses
  Interventions: Diagnostic Test: The Quality of Vision questionnaire
- AcrySof IQ PanOptix intraocular lenses: Eyes of patients undergoing cataract surgery with implantation of AcrySof IQ PanOptix (Alcon Laboratories, Inc.) intraocular lenses
  Interventions: Diagnostic Test: The Quality of Vision questionnaire

INTERVENTIONS:
Diagnostic Test: The Quality of Vision questionnaire — The Quality of Vision questionnaire rates glare, halos, starbursts, hazy/blurred/double vision, distortion, focusing difficulties, fluctuation, and depth perception conditions.

SUMMARY:
The purpose of the present study was to compare the clinical outcomes such as visual function, refraction errors and visual quality of patients undergoing cataract surgery with implantation of two different models of diffractive trifocal IOLs: RayOne Trifocal (Rayner IOL, Ltd.) and AcrySof IQ PanOptix (Alcon Laboratories, Inc.) IOL.

DETAILED DESCRIPTION:
Cataract is affecting over 95 million people worldwide and remains the leading cause of vision impairment and blindness. Cataract surgery is an effective method for restoring visual acuity (VA). With the advancement of cataract surgery technique and intraocular lenses (IOL) technologies, expectations of patients from cataract surgery have good vision at distance and near ranges without using spectacles. The standard IOLs design were monofocal, which offered only fixed focal distance. One of the main factors for dissatisfaction after monofocal pseudophakic eyes is lack of accommodation. Previous studies demonstrated that this problem can be resolved by using diffractive trifocal IOLs. Diffractive trifocal IOLs provide effective near, intermediate and distance visual restoration, and has been widely used in patients who want to achieve spectacle independence after surgery. However, some possible optical side effects of trifocal IOLs have been reported, including halos and other dysphotopsias, reduced contrast sensitivity (CS), glare disability, which can significantly affect visual quality and patient satisfaction. The purpose of the present study was to compare the clinical outcomes such as visual function, refraction errors and visual quality of patients undergoing cataract surgery with implantation of two different models of diffractive trifocal IOLs: RayOne Trifocal (Rayner IOL, Ltd.) and AcrySof IQ PanOptix (Alcon Laboratories, Inc.) IOL.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent cataract surgery with trifocal intraocular lenses implantation in one or both eyes

Exclusion Criteria:

* Amblyopia
* Axial length (AL) over 25 mm
* Previous history of corneal or refractive surgery
* Ocular comorbidity (corneal scars, keratoconus, and corneal endothelial dystrophy, chronic or recurrent uveitis, macular degeneration, diabetes mellitus with retinal changes, glaucoma or intraocular pressure equal or higher than 24 mmHg)
* Patient inability to understand and/or fill in patient questionnaires

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients underwent cataract surgery with trifocal intraocular lenses implantation in one or both eyes at Akdeniz University Hospital Ophtalmology Department.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
The Quality of Vision score | 3 months
  Glare, halos, starbursts, hazy/blurred/double vision, distortion, focusing difficulties, fluctuation, and depth perception

CONTACTS AND LOCATIONS:
Locations (1):
- Aslı Çentinkaya Yaprak, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No